CLINICAL TRIAL: NCT04405401
Title: Stereotactic Ablative Radiotherapy for Oligo-Progressive Disease REfractory to Systemic Therapy in Non Small Cell Lung Cancer: A Registry-based Phase II Randomized Trial
Brief Title: Stereotactic Ablative Radiotherapy for Oligo-Progressive Non Small Cell Lung Cancer
Acronym: SUPPRESS-NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-9066
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer Metastatic
Keywords: non small cell lung cancer; oligoprogression; steretactic body radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized screening phase II trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Switch to subsequent systemic therapy line, best supportive care or continue current systemic line
  Interventions: Radiation: SABR
- Experimental SABR arm (Experimental): Definitive SABR to oligoprogressive lesions + continue current systemic therapy
  Interventions: Other: Standard of care

INTERVENTIONS:
Radiation: SABR — SABR to all oligoprogressive lesions + continuation of current systemic therapy
  Arms: Standard of care
Other: Standard of care — Patients on the standard arm will be treated as per standard of care in our institution. Treatment options could include switching to next systemic therapy line, best supportive care or continuing on current systemic therapy.
  Arms: Experimental SABR arm

SUMMARY:
A registry-based randomized screening phase II trial. A total of 68 patients with metastatic non small cell lung cancer on systemic therapy with oligoprogression to 1-5 extracranial lesions will be randomized using a 1:1 ratio to standard of care (begin next-line systemic therapy, best supportive care, continue current systemic line, based on treating physician decision) vs. receive stereotactic ablative radiotherapy to all oligoprogressive lesions while continuing their current systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Metastatic NSCLC enrolled in our CRCHUM Lung Cancer Registry and co-enrolled to the PERa registry
* Ability to provide written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* Oligoprogression to 1-5 extracranial lesions ≤ 5cm and involving ≤ 3 organs. Progression at the primary tumor site should be counted within the total of 5 lesions. For patients with lymph node metastases, each node is counted as one site of metastasis.
* Oligoprogression while on ICI or TKI (any line)
* Patients with brain metastasis are allowed; brain metastasis are not counted in the maximum number of lesions and should be treated as per standard of care
* All sites of disease can, in the opinion of the investigator, be safely treated and targetable with SABR (taking into account prior local therapy, organ function and underlying medical condition such as inflammatory bowel disease, pulmonary fibrosis, etc.)
* Patients with prior metastases that have been treated with ablative therapies (e.g. radiotherapy, surgery or radiofrequency ablation) before their current line of systemic therapy, are eligible.

Exclusion Criteria:

* Any lesion beyond 5 cm
* Pregnancy or breastfeeding
* Any medical condition that could, in the opinion of the investigator, preclude radiotherapy or prevent follow-up after radiotherapy.
* Presence of spinal cord compression Metastatic disease that invades the GI tract (including esophagus, stomach, small or large bowel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 5 years
  PFS defined from randomization to disease progression at any site or death
OS | 5 years
  OS defined as time from randomization to time of death from any cause.

SECONDARY OUTCOMES:
Quality of life Measured using the FACT-G tool, lung cancer-related patient reported outcome- CTCAE (PRO-CTCAE) | 5 years
  Measured using the FACT-G tool, lung cancer-related patient reported outcome- CTCAE (PRO-CTCAE)
Quality of life 5-level EQ-5D (EQ-5D-5L) | 5 years
  questionnaire
Grade ≥ 3 toxicity | 5 years
  Measured using the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Local control | 5 years
  Defined as time from the end of SABR treatment to date of local failure and will be measured only in the experimental arm
Time to next systemic therapy | 5 years
  Defined as time from randomization to time of subsequent therapy line

CONTACTS AND LOCATIONS:
Overall Officials: Houda Bahig, MD PhD, Study Chair — Centre hospitalier de l'Université de Montréal (CHUM); Bertrand Routy, MD PhD, Study Chair — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided